CLINICAL TRIAL: NCT02150616
Title: Patients With Pulmonary Hypertension or Interstitial Lung Disease Travelling to Altitude - Effect of Nocturnal Oxygen Therapy on Breathing and Sleep
Brief Title: Patients With Pulmonary Hypertension or Interstitial Lung Disease at Altitude - Effect of Oxygen on Breathing and Sleep
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ID 2013-0088V2A3D
Record Dates: First submitted 2014-05-18; First posted 2014-05-30 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-01

CONDITIONS: Precapillary Pulmonary Hypertension; Interstitial Lung Disease
Keywords: Pulmonary hypertension; Interstitial lung disease; Pulmonary fibrosis
MeSH Terms: conditions — Lung Diseases, Interstitial; Hypertension, Pulmonary; Pulmonary Fibrosis | interventions — WW Domain-Containing Oxidoreductase; Oxygen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Moderate altitude sojourn (Experimental): Sojourn at moderate altitude (2048 m)
  Interventions: Behavioral: Moderate altitude sojourn; Behavioral: Low altitude sojourn; Drug: Oxygen; Drug: Sham oxygen (room air)
- Low altitude sojourn (Experimental): Sojourn at low altitude (490 m, baseline)
  Interventions: Behavioral: Moderate altitude sojourn; Behavioral: Low altitude sojourn; Drug: Oxygen; Drug: Sham oxygen (room air)
- Oxygen (Active Comparator): Oxygen administration via a nasal cannula at a rate of 3 L/min during nights spent at 2048 m
  Interventions: Behavioral: Moderate altitude sojourn; Behavioral: Low altitude sojourn; Drug: Oxygen; Drug: Sham oxygen (room air)
- Sham oxygen (room air) (Placebo Comparator): Sham oxygen (room air) administration via a nasal cannula at a rate of 3 L/min during nights
  Interventions: Behavioral: Moderate altitude sojourn; Behavioral: Low altitude sojourn; Drug: Oxygen; Drug: Sham oxygen (room air)

INTERVENTIONS:
Behavioral: Moderate altitude sojourn — Participants will travel from Zurich (490 m) to St. Moritz Salastrains (2048 m) and stay there for 2 days
  Other Names: Moderate altitude sojourn at 2048 m for 2 days
Behavioral: Low altitude sojourn — Low altitude baseline evaluations will be performed during a stay at Zurich (490)
  Other Names: Low altitude sojourn at 490 m (Zurich) for 1.5 days
Drug: Oxygen — Oxygen administration via a nasal cannula at a rate of 3 L/min during nights spent at 2048 m
  Other Names: Nocturnal nasal oxygen administration during stay at 2048 m
Drug: Sham oxygen (room air) — Sham oxygen (room air) administration via a nasal cannula at a rate of 3 L/min during nights at 490 m and 2048 m
  Other Names: Nocturnal nasal room air administration

SUMMARY:
The purpose of this study is to investigate the effect of travelling to moderate altitude and of nocturnal oxygen therapy during a stay at moderate altitude on breathing and sleep of patients with pulmonary hypertension or with interstitial lung disease.

DETAILED DESCRIPTION:
Patients with pulmonary hypertension or with interstitial lung disease living below 800 m will be invited to participate in a randomized, cross-over field trial evaluating the hypotheses that: a), breathing and sleep during a 2 day sojourn at moderate altitude are impaired in comparison to low altitude; b), breathing and sleep during a 2 day sojourn at moderate altitude are improved by nocturnal oxygen therapy compared to room air (sham oxygen) administered during nights at altitude. Outcomes will be assessed at low altitude (Zurich, 490 m, baseline), and during 2 study periods of 2 days each spent at moderate altitude (St. Moritz Salastrains, 2048 m), separated by a wash-out period of at least 2 weeks spent at low altitude (<800 m). The order of stays at the different altitudes and of the treatments will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Precapillary pulmonary hypertension, or interstitial lung disease.
* New York Heart Association class 2-3.
* Residence at low altitude (<800m).

Exclusion Criteria:

* Unstable or exacerbated condition
* Very severe pulmonary hypertension or interstitial lung disease, New York Heart Association class 4
* requirement for oxygen therapy at low altitude residence
* hypoventilation
* more than mild or unstable cardiovascular disease
* use of drugs that affect respiratory center drive
* internal, neurologic or psychiatric disease that interfere with protocol compliance including current heavy smoking (>20 cigarettes per day), inability to perform 6 min walk test.
* previous intolerance to moderate altitude (<2600m).
* Exposure to altitudes >1500m for >2 days within the last 4 weeks before the study.
* Pregnant or nursing patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-05; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Mean nocturnal oxygen saturation measured by pulse oximetry | Approximately 8 hours (during the first night at 2048 m)
  Difference in mean nocturnal oxygen saturation between measurements at 2048 m (altitude) and 490 m (baseline); and between the oxygen and sham oxygen treatment periods at 2048 m.
Apnea/hypopnea index measured by polysomnography | Approximately 8 hours (during the first night at 2048 m)
  Difference in apnea/hypopnea index between measurements at 2048 m (altitude) and 490 m (baseline); and between the oxygen and sham oxygen treatment periods at 2048 m.

SECONDARY OUTCOMES:
Mean nocturnal oxygen saturation measured by pulse oximetry | Approximately 8 hours (during the second night at 2048 m)
  Difference in mean nocturnal oxygen saturation between measurements at 2048 m (altitude) and 490 m (baseline); and between the oxygen and sham oxygen treatment periods at 2048 m.
Apnea/hypopnea index measured by polygraphy | Approximately 8 hours (during the second night at 2048 m)
  Difference in apnea/hypopnea index between measurements at 2048 m (altitude) and 490 m (baseline); and between the oxygen and sham oxygen treatment periods at 2048 m.
Sleep quality visual analog scale score | Approximately 8 hours (during the first night at 2048 m)
  Difference in subjective sleep quality between visual analog scale measurements at 2048 m (altitude) and 490 m (baseline); and between the oxygen and sham oxygen treatment periods at 2048 m.
Psychomotor vigilance test reaction time | Approximately at 10 a.m. on the second day at 2048 m
  Difference in reaction time between measurements at 2048 m (altitude) and 490 m (baseline); and between the oxygen and sham oxygen treatment periods at 2048 m.
Severe hypoxemia | Approximately 72 hours, Day 1 to 3 at 2048 m
  Number of participants in whom arterial oxygen saturation measured by pulse oximetry is less than 75% for more than 30 min during the sojourn at 2048 m (altitude) and 490 m (baseline); and during the oxygen and sham oxygen treatment periods at 2048 m.
Subjective sleep quality visual analog scale score | Approximately 8 hours (during the second night at 2048 m)
  Difference in subjective sleep quality between visual analog scale measurements at 2048 m (altitude) and 490 m (baseline); and between the oxygen and sham oxygen treatment periods at 2048 m.

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Study Chair — University Hospital, Zürich
Locations (1):
- University Hospital Zurich, Pulmonary Division, Zurich, Switzerland